CLINICAL TRIAL: NCT04231760
Title: The Effect of Inhaled Nitric Oxide on Pulmonary Gas-exchange in COPD
Acronym: iNO
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: Pro00092368
Record Dates: First submitted 2020-01-14; First posted 2020-01-18 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Chronic Obstructive Pulmonary Disease (Experimental): Mild & Moderate COPD to receive either placebo or inhaled nitric oxide (40ppm)
  Interventions: Drug: Inhaled Nitric Oxide; Drug: Placebo
- Healthy Controls (Active Comparator): Control group to receive either placebo or inhaled nitric oxide (40ppm)
  Interventions: Drug: Inhaled Nitric Oxide; Drug: Placebo

INTERVENTIONS:
Drug: Inhaled Nitric Oxide — Inhaled nitric oxide, which consists of breathing medical grade air (21% O2) with 40 parts per million of nitric oxide.
Drug: Placebo — Inhaled placebo, which consists of breathing medical grade air (21% O2).

SUMMARY:
Chronic Obstructive Pulmonary Disease (COPD) is a lung disorder commonly caused by smoking, which makes breathing more difficult. When COPD patients exercise, they are not efficient breathers and this leads to serious breathing difficulties, which often causes these patients to stop exercise at low intensities. Even though patients with a mild form of COPD have relatively well preserved lung function, they still have inefficient breathing during exercise. The investigators think that these individuals have problems exchanging fresh gas (i.e., oxygen) into the blood stream because of poor lung blood vessel function. The investigators will test whether inhaled medications, specifically nitric oxide, can improve lung blood vessel function and decrease breathing difficulties during exercise. With this research, the investigators will understand more about breathing efficiency and lung blood vessel function in individuals with mild COPD, and find out whether improving lung blood vessel function helps COPD patients breathe easier and exercise longer. Understanding the reasons behind the feeling of difficult breathing may lead to more effective therapy and improved quality of life in COPD patients.

DETAILED DESCRIPTION:
BACKGROUND

Chronic Obstructive Pulmonary Disease (COPD) is a respiratory disorder typically caused by smoking and is characterized by airway obstruction. Exertional dyspnea (perceived breathlessness) is a hallmark of COPD regardless of severity and is the primary reason for exercise intolerance even in patients with mild COPD. Dyspnea in COPD has been shown to profoundly reduce patient quality of life, physical activity, and impair patients' ability to complete day-to-day tasks. Previous work in mild COPD has demonstrated that exertional dyspnea is the result of increased work of breathing during exercise, and that this increased work of breathing comes from: 1) an exaggerated ventilatory response to exercise (i.e. increased minute ventilation relative to carbon dioxide production, V̇E/V̇CO2), and 2) airflow limitation (i.e. expiratory flow limitation and resulting dynamic hyperinflation). A great deal of work has focused on improving airflow limitation in COPD; however, very little has been done to understand and treat the exaggerated ventilatory response to exercise in COPD.

Several previous studies in mild COPD have consistently shown an elevated ventilatory response (i.e. greater V̇E/V̇CO2) during exercise. The elevated V̇E/V̇CO2 response to exercise appears to be clinically important, as it independently predicts mortality in COPD. This increased V̇E/V̇CO2 in mild COPD appears to be secondary to increased deadspace ventilation (i.e. sections of the lung with ventilation, but no perfusion), and this increased deadspace ventilation results in a compensatory increase in total minute ventilation (i.e. increased V̇E/V̇CO2) to maintain effective alveolar ventilation and arterial blood gas homeostasis.

The underlying mechanism(s) for the increased deadspace ventilation and V̇E/V̇CO2 during exercise in mild COPD is currently unclear; however, pulmonary microvascular abnormalities and hypoperfusion of pulmonary capillaries are potential pathophysiologic mechanisms. Downregulation of NO bioavailability, secondary to persistently reduced endothelial NO synthase (eNOS), contributes to pulmonary vascular endothelial dysfunction and the development of both emphysema and pulmonary arterial hypertension (PAH) in COPD. Inhaled nitric oxide (iNO) is used to treat disorders of the pulmonary vasculature such as forms of PAH. By increasing NO bioavailability, pulmonary vascular function is improved. Previous work in PAH patients has shown that typical clinical doses (20-40 parts per million (ppm)) of iNO can reduce pulmonary vascular resistance and increase exercise capacity (V̇O2peak). Despite emerging evidence that COPD is associated with pulmonary vascular dysfunction, there is limited research investigating iNO as a therapeutic intervention in COPD. The investigators recently completed a randomized double-blinded controlled trial examining the effectiveness of 40 ppm iNO on V̇O2peak in mild COPD. As compared to placebo (inhaled room air), iNO improved V̇O2peak and dyspnea in COPD secondary to a reduction in ventilatory inefficiency (V̇E/V̇CO2), suggesting that vascular dysfunction is an important contributor to ventilation, dyspnea and exercise intolerance in mild COPD.

The reduction in V̇E/V̇CO2 during exercise with iNO would suggest that iNO increases pulmonary microvascular perfusion, leading to improved V̇A/Q̇ matching, reduced deadspace ventilation and therefore reduced ventilation for a given metabolic demand. However, this needs to be demonstrated experimentally. The gold standard for evaluation of V̇A/Q̇ matching is the multiple inert gas elimination technique (MIGET), as this technique is able to quantify V̇A/Q̇ matching by the relative distribution of ventilation (log SDV) and perfusion (log SDQ)27. Further, MIGET allows for quantification of pure deadspace (sections of ventilation with no perfusion) as compared to high V̇A/Q̇ regions of the lung (i.e. ventilation with low relative perfusion). Should iNO reduce deadspace and improve V̇A/Q̇, this would clearly establish that vascular dysfunction (and not vascular destruction) contributes to V̇A/Q̇ mismatch in mild COPD, and that the reduction in V̇E/V̇CO2 and improvement in exercise capacity with iNO is explained by improved V̇A/Q̇ matching. Further, this finding would help identify a vascular target to improve dyspnea, exercise tolerance, and by extension quality of life in COPD.

STUDY PURPOSE AND DESIGN

Purpose: To determine the effect of iNO on ventilatory demand and V̇A/Q̇ matching during exercise in individuals with COPD.

Hypothesis: Inhaled NO will reduce ventilatory demand during exercise, secondary to improved V̇A/Q̇ matching during exercise in individuals with COPD.

Study Design: Randomized double-blind cross-over design.

Study Protocol: Four sessions will be completed over a 4-week period in the following order:

Day 1): Participant enrollment, medical history, standard pulmonary function and cardiopulmonary exercise test (CPET). Day 2): Resting cardiac ultrasound. Day 3): Participants will complete two separate experimental conditions breathing either room air (placebo, 21% O2, 79% N2) or iNO (room air with 40 ppm NO). The order of condition will be randomized using a concealed randomized methodology, and the participant will breathe through the identical apparatus throughout both conditions. Within each condition, data will be gathered at 3 stages: 1) in the resting upright position, 2) during exercise at 30% of V̇O2peak, and 2) at the exercise intensity corresponding to their nadir V̇E/V̇CO2 (workload determined during CPET, and typically ~60% V̇O2peak). All physiological measurements will be completed at each stage. A 15 minute break between each condition will be given to allow for recovery and washout of NO. Day 4): Participants will repeat the exercise protocol as described in Day 3, however, only MIGET data will obtained while operating lung volume data will not be gathered so as to ensure high-quality MIGET data. Each visit will take approximately 3 hours. The total time duration for each participant will be approximately 12 hours.

On Day 1, participants will complete the informed consent procedure and be screened for exercise using a medical history questionnaire. They will undergo lung function, resting echocardiography and cardiopulmonary exercise testing on the same day. The participants will be spending approximately three hours in the laboratory on this testing day.

On Day2, the participant will lie in a semi-supine and be rested for 5 minutes. There cardiac function and pulmonary arterial systolic pressure will then be measured using echocardiography. Measurements will be made while the participants breathing breathe medical grade air (room air) or room air titrated with 40 parts per million of nitric oxide

On days 3 & 4 (one day per week in 2 consecutive weeks), the participants will breathe medical grade air (room air) or room air titrated with 40 parts per million of nitric oxide and have their blood flow/cardiac output, arterial blood gas and expired gas evaluated during sub-maximal exercise. The participants will complete both conditions (room air & nitric oxide) on each day, in random order.

On day 3, the participant will lie supine and be rested for 5 minutes. Their resting blood pressure will be determined using manual auscultation. Resting cardiac output will be evaluated using noninvasive impedance cardiography and oxygen saturation estimated with pulse oximetry. Ventilation will be measured from expired gas analysis. Following these measurements, the participant will begin to breathe medical grade room air. Following a 20 minute wash-in period, ventilation, cardiac output and oxygen saturation recordings will be repeated. Participants will then exercise on a cycle ergometer while continuing to breathe the medical grade room air and all physiological measurements will be repeated. After a short break (minimum 15 minutes), the 20-minute wash in and exercise bout will be repeated in the nitric oxide condition. The participants will be spending approximately three hours in the laboratory on this testing day.

Day 4 will be identical to day 3 except, however, arterial blood gas will also be sampled at rest and during exercise. Further, a venous catheter will be inserted into the ante-cubital vein and a solution containing 6 inert gases will be infused to allow assessment of ventilation-perfusion matching using the multiple inert gas elimination technique (MIGET). The arterial and venous catheter will be inserted by either a certified cardiologist or respirologist. Further details regarding catheterization and MIGET are detailed below in the outcomes section.

Intervention

Inhaled Nitric Oxide Intervention: Inhaled NO is a selective pulmonary vasodilator and has been shown to improve blood flow to well-ventilated lung areas (i.e. improve V̇A/Q̇ matching) in conditions with elevated vascular tone. Inhaled NO has been previously shown to lower pulmonary artery pressure during exercise in severe COPD patients, while not affecting systemic blood pressure. It is important to note that a selective pulmonary vasodilator will be used instead of an intravenously infused vasodilator (e.g. prostacyclin) to avoid systemic vasodilation, severe arterial hypotension and syncope. Consistent with previous work, a standard 40 ppm dose of inhaled NO will be administered using a non-rebreathing circuit.

Statistical analysis and Interpretation: Unpaired t-analysis will be used to compare demographics between the COPD group and the controls. A mixed effects linear regression model will be used to evaluate changes in V̇A/Q̇ inequality, specifically the variability in perfusion (log SDQ, primary outcome), with the intervention. Fixed effects will be intervention (placebo vs. iNO), workload (rest, 30% V̇O2peak, power output at nadir V̇E/V̇CO2), period (i.e. randomization order) and random effects will represent participants and intervention order. Sex will also be included in the model as well as interactions. Similar models will be developed for each secondary outcome (log SDV, deadspace ventilation, V̇E/V̇CO2). Hypotheses and other aspects (e.g. carry-over effect) will be assessed by testing various contrasts.

ELIGIBILITY:
Inclusion Criteria:

* Twenty participants with mild COPD (forced expiratory volume in 1 s (FEV1)/forced vital capacity (FVC) below the lower limit of normal (<-1.64 z-score)1) and FEV1 ≥ 80% predicted, with a smoking history (10 > pack-years) will be recruited. Twenty participants with moderate COPD (FEV1/ FVC below the lower limit of normal (<-1.64 z-score)1) and FEV1 50-80% predicted, with a smoking history (10 > pack-years) will also be recruited. Additionally, 40 healthy individuals with be recruited.
* Participants will be free of any known significant cardiovascular, metabolic or neuromuscular disease. Participants with COPD will have global initiative for chronic obstructive lung disease (GOLD) Stage 1 mild COPD (FEV1/FVC ratio <0.70 and FEV1 ≥ 80% predicted1) and Stage 2 moderate COPD (FEV1/FVC ratio <0.70 and FEV1 50-80% predicted) and a >10 pack-year smoking history. Controls will have normal lung function, minimal smoking history and no previous diagnosis of COPD. Participants will range from 18-85 years old.

Exclusion Criteria:

* Individuals with significant cardiovascular, metabolic, neuromuscular or any other disease that could contribute to dyspnea or abnormal cardiopulmonary responses to exercise will be excluded.
* Individuals with musculoskeletal injuries that prevent them from completing cycle ergometry exercise trials will be excluded.
* COPD participants currently on oral steroids (i.e. prednisone), phosphodiesterase type 5 (PDE5) inhibitors or supplemental O2 therapy will be excluded.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2026-12-01 (Estimated); Primary Completion 2027-12-01 (Estimated); Study Completion 2028-02-01 (Estimated)

PRIMARY OUTCOMES:
Ventilation-perfusion matching | Within 20-25 minutes post-dose
  Using the multiple inert gas elimination technique, ventilation-perfusion matching at rest and during exercise will be quantified by the second moment perfusion distribution (log standard deviation of the perfusion distribution (log SDQ)).

SECONDARY OUTCOMES:
Ventilation | Within 20-25 minutes post-dose
  Ventilatory response at rest and during exercise quantified using expired gas analysis

CONTACTS AND LOCATIONS:
Overall Officials: Michael Stickland, PhD, Principal Investigator — University of Alberta

IPD SHARING:
Plan to Share IPD: No